CLINICAL TRIAL: NCT00151567
Title: Interest of a Treatment With the alpha1-blocker Tamsulosin in the Elimination of Pelvis Ureteral Stones
Brief Title: Evaluation of Tamsulosin in the Treatment of Ureteral Stones
Acronym: TAMSULOSINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government); Yamanouchi (Unknown)
Responsible Party: Direction of Clinical Research, Rennes University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFSSAPS 010751; PHRC/00-01 (Other: Rennes University Hospital); CIC0203/004
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2008-09

CONDITIONS: Ureterolithiasis; Ureteral Calculi
Keywords: Ureterolithiasis; Alpha1-blocker; Lower ureteral stone
MeSH Terms: conditions — Ureterolithiasis; Ureteral Calculi | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Tamsulosin
  Interventions: Drug: Tamsulosin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamsulosin — Oral tamsulosin once a day until stone elimination or the end of the follow-up (42 days)
  Arms: 1
Drug: Placebo — Oral placebo of tamsulosin once a day until stone elimination or the end of the follow-up (42 days)
  Arms: 2

SUMMARY:
Ureteral stones have an important place in daily urological practice, usually causing acute episodes of ureteral colic by obstructing the urinary tract. The aim of the study is to evaluate whether repeated administration of tamsulosin, a drug routinely used in the treatment of lower urinary tract symptoms, could lower the delay of elimination of the stone in patients with pelvis ureterolithiasis.

DETAILED DESCRIPTION:
Ureteral colic, mainly due to ureterolithiasis, represents 1 to 2% of hospital emergency admissions. When a surgical intervention is not required, usual treatment combines hydration and anti-inflammatory drugs.

Alpha1-blockers, firstly developed as anti-hypertensive drugs, are now also used in the management of benign prostatic hyperplasia, due to their relaxing properties on the urinary tract. The aim of the study is to investigate whether tamsulosin could lower the delay of elimination of the stone in patients with pelvis ureterolithiasis. Patients are randomized to receive either tamsulosin or a placebo in addition to usual treatment until stone elimination. Efficacy is assessed by evaluating the time to spontaneous passage of the stone between day 1 and day 42, the need for surgery and pain recurrences.

ELIGIBILITY:
Inclusion Criteria:

* Adult over 18 years
* Emergency admission for a ureteral colic
* Radio-opaque ureterolithiasis
* Stone of 2 to 7 mm diameter
* Informed written consent

Exclusion Criteria:

* Pregnancy or breast-feeding
* Treatment with alpha or beta-blocker
* Contraindication to tamsulosin (orthostatic hypertension, hepatic failure)
* Complication needing surgery
* Calculi spontaneous passage before randomization
* Patient not available for a 6 week follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2002-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Time to stone elimination in days (censored criterion) | between day 1 and 42

SECONDARY OUTCOMES:
Time to stone elimination in days in patients with spontaneous elimination (quantitative criterion) | between day 1 and 42
Pain using Visual Analogue Scale | days 1, 2, 3
Spontaneous stone elimination rate | days 1, 7, 14, 21, 28, 35, and 42
Spontaneous stone elimination rate, according to stone size (2-3 mm, 4-5 mm, 6-7 mm) | days 1, 7, 14, 21, 28, 35, and 42
Rate of need for surgery | Within 42 days
Time to surgery in days in patients with surgical elimination | between day 1 and day 42
Rate of pain recurrences | within 42 days
Time to the first recurrence in days | between day 1 and day 42
Rate of need for corticoids or morphine | Within 42 days
Time to the first administration of corticoids or morphine in days | between day 1 and day 42
Rate of adverse events | Within 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Francois Guillé, MD, Principal Investigator — Rennes University Hospital; Eric Bellissant, MD, PhD, Study Chair — Rennes University Hospital
Locations (6):
- France (6):
  - Service d'Urologie- Hôpital du Val de Grâce, Paris
  - Service d'Urologie - Hôpital de La Milétrie, Poitiers
  - Hôpital de Redon, Redon
  - Service d'Urologie- Hôpital Robert Debré, Reims
  - Service d'Urologie- Hôpital Pontchaillou, Rennes
  - Service d'Urologie - Hôpital Bretonneau, Tours

REFERENCES:
- [Background] Resim S, Ekerbicer H, Ciftci A. Effect of tamsulosin on the number and intensity of ureteral colic in patients with lower ureteral calculus. Int J Urol. 2005 Jul;12(7):615-20. doi: 10.1111/j.1442-2042.2005.01116.x. PMID 16045553
- [Background] Wilde MI, McTavish D. Tamsulosin. A review of its pharmacological properties and therapeutic potential in the management of symptomatic benign prostatic hyperplasia. Drugs. 1996 Dec;52(6):883-98. doi: 10.2165/00003495-199652060-00012. PMID 8957159
- [Derived] Vincendeau S, Bellissant E, Houlgatte A, Dore B, Bruyere F, Renault A, Mouchel C, Bensalah K, Guille F; Tamsulosin Study Group. Tamsulosin hydrochloride vs placebo for management of distal ureteral stones: a multicentric, randomized, double-blind trial. Arch Intern Med. 2010 Dec 13;170(22):2021-7. doi: 10.1001/archinternmed.2010.447. PMID 21149761